CLINICAL TRIAL: NCT01153100
Title: Effectiveness of a Subcutaneously Administered Long-acting Insulin Added to Insulin Drip Therapy as Compared With Standard Insulin Drip Treatment
Brief Title: Effectiveness of Adding Subcutaneous Long-acting Glargine to Insulin Drip Therapy Compared With Standard Insulin Drip Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-1065
Record Dates: First submitted 2010-06-14; First posted 2010-06-29 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard insulin drip therapy (No Intervention): Standard insulin drip therapy
- Insulin drip and glargine (Active Comparator): Insulin drip and glargine 0.25 units per kg body weight
  Interventions: Drug: Glargine

INTERVENTIONS:
Drug: Glargine — Glargine 0.25 units per kg body weight given every 24 hours while patients are receiving intravenous (IV) standard insulin drip therapy
  Other Names: Lantus
  Arms: Insulin drip and glargine

SUMMARY:
The investigators anticipate that the use of Glargine will decrease the duration of an insulin drip, the dose of short-acting insulin in the drip, hospital and ICU (intensive care unit) length of stay, improve glycemic control, and prevent rebound hyperglycemias when the insulin drip is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic ketoacidosis (DKA) and hyperglycemic hyperosmolar non-ketotic states, hyperglycemia with severe illness, pre- and postoperative states, nothing by mouth (NPO), as well as gastric (tube feeding) and parenteral nutrition requiring insulin drip.
* Patients with type 1 and type 2 diabetes mellitus (DM) will be included.
* Patients with both types of diabetes will be among those treated with the insulin drip while being NPO, having severe concomitant illness or receiving enteral and parenteral nutrition.
* Patients will be of age 19 to 80.

Exclusion Criteria:

* Inability to consent for the study for any reason including cognitive impairment secondary to hyperglycemia, presence of severe medical conditions requiring intubation, severe sepsis, hypothermia, and anticipated length of insulin drip 2 weeks and longer, pregnancy, Lantus allergy, and concurrent sulfonamide treatment

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Reduction in rebound hyperglycemia (blood glucose levels over 180 mg/dl) | within 48 hours of discontinuation

SECONDARY OUTCOMES:
Reduction in duration of insulin drip therapy and reduction in total and average per hour insulin drip dose | within one week of insulin drip therapy
Reduction in ICU length of stay | within two weeks of hospitalization
Equal or improved diabetes control | within two weeks of hospitalization
Reduction in time to get back to control of glycemia (140-180 mg/dl) if rebound hyperglycemia occurs | within one week post insulin drip

CONTACTS AND LOCATIONS:
Overall Officials: Boris Draznin, MD, Principal Investigator — Univesity of Colorado
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States